CLINICAL TRIAL: NCT05703386
Title: Imaging the Pathogenesis of Cerebral Small Vessel Disease
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00313202
Record Dates: First submitted 2023-01-06; First posted 2023-01-30 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Ischemic Stroke; Hypertension; Hyperlipidemias; Diabetes
Keywords: Cerebral small vessel disease; Vascular cognitive impairment and dementia; White matter hyperintensities; Blood-brain barrier; Vascular risk factors; Ischemic stroke
MeSH Terms: conditions — Ischemic Stroke; Hypertension; Hyperlipidemias; Diabetes Mellitus; Cerebral Small Vessel Diseases; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cerebral small vessel disease (CSVD) can lead to vascular cognitive impairment and dementia (VCID). The hallmark of CSVD is the appearance and progression of white matter hyperintensities (WMH) on MRI. The goal of this study it to recruit and follow individuals at risk for WMH progression and use serial MRI scanning to gain insights into the pathogenesis of CSVD.

DETAILED DESCRIPTION:
Vascular Cognitive Impairment and Dementia (VCID) which is attributed in large part to cerebral small vessel disease (CSVD) is prevalent in patients with a history of stroke and vascular risk factors. The hallmark of CSVD is white matter hyperintensities (WMH) seen on T2-weighted MRI. The initial amount, and rate of progression, of WMH is tied closely with the development and progression cognitive deficits. It is hypothesized that one of the early pathologic features in the normal appearing white matter (NAWM), before it progresses to WMH is disruption of the blood-brain barrier (BBB) and loss of micro-structural integrity. The purpose of this study is track the progression of WMH using multiple MRI biomarkers looking at BBB disruption (DCE, DSC, ASL), micro-structural changes (multi-shell DTI), and macrostructural changes (FLAIR, SWI, T1) to better understand the pathogenesis of CSVD. Patients with a history of a stroke, at least one vascular risk factor, and evidence of CSVD on MRI may be eligible for this study. We will follow 50 patients with 3 MRIs performed over 1.25 years

ELIGIBILITY:
Inclusion Criteria:

* Clinical or radiographic evidence of ischemic stroke
* One vascular risk factor (hypertension, hyperlipidemia, or diabetes)
* Evidence of cerebral small vessel disease on MRI

Exclusion Criteria:

* Inability to complete 3 research MRI scans over 1.25 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who are identified as having had an ischemic stroke, have at least one vascular risk factor, have had an MRI demonstrating cerebral small vessel disease and are willing and able to come to our research facility in Baltimore for 3 MRI scans over 1.25 years.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-11-08 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Progression of cerebral small vessel disease | 1 year
  Conversion of normal appearing white matter to white matter hyperintensity measured on MRI using 3D FLAIR imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Leigh, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided